CLINICAL TRIAL: NCT06413134
Title: A Prospective, Randomized, Crossover Study of Therapy Adherence With TheraPAP Compared to Automatic Adjusting Positive Airway Pressure (APAP) for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: TheraPAP Adherence Crossover Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This was supposed to be a pilot, single center study, which has been de-prioritized. A larger study will be conducted instead
Sponsor: SleepRes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Home 0001
Record Dates: First submitted 2024-05-03; First posted 2024-05-14 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: There will be two, 6-week arms where patients will breathe on standard APAP therapy and the test therapy, TheraPAP. Starting therapy will be randomly assigned, but all participants will sleep using both therapies.
Who Masked: Participant
Masking Description: Participants will not be told what therapy they will be using in either arm, and since they are naive to PAP therapy, they would be more blinded than adherent patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 6-weeks breathing on APAP (Placebo Comparator): Patients will breathe on APAP for 6 weeks simulating normal therapy. Usage, leak, P95/P90 and AHI will be recorded and averaged over the duration.
  Interventions: Device: APAP
- 6-weeks breathing on TheraPAP (Experimental): Patients will breathe on TheraPAP for 6 weeks, which is the therapy under evaluation. Usage, leak, P95/P90 and AHI will also be recorded and averaged over the duration.
  Interventions: Device: TheraPAP

INTERVENTIONS:
Device: TheraPAP — TheraPAP is a novel CPAP-based therapy in which pressure is dropped as much as 5 cmH2O starting at the beginning of inspiration and extending through the end of expiration where it rises back up to the true therapy pressure for a short period. It improves comfort by providing pressure only when it is needed and maintaining it at a low level the rest of the time. Normal CPAP/APAP therapy keeps pressure at the therapy level during the entire breath cycle, except with some alternate approaches where pressure is decreased but only during the expiratory phase.
  Other Names: KPAP
  Arms: 6-weeks breathing on TheraPAP
Device: APAP — Standard CPAP therapy where therapy pressure is automatically adjusted to prevent respiratory events from occurring. The TheraPAP prototype device will be used to operate in the APAP mode in addition to the TheraPAP intervention mode.
  Arms: 6-weeks breathing on APAP

SUMMARY:
TheraPAP is a novel therapy approach being developed by SleepRes, LLC. for the treatment of obstructive sleep apnea (OSA). This algorithm has been integrated into the Sefam S.Box CPAP (continuous positive airway pressure) device and both standard CPAP/APAP (auto-titrated PAP) as well as TheraPAP can be delivered. TheraPAP is a pressure control algorithm that lowers the pressure from the set pressure at the beginning of inspiration and does not return the pressure to the full set level until some point in late expiration. In this randomized crossover study, the comparative adherence to therapy between TheraPAP and APAP will be compared. Each therapy will be used by the patient for six-week periods with randomly assigned order, and the usage during each arm will be compared.

DETAILED DESCRIPTION:
The TheraPAP Adherence Study is a randomized, crossover study in treatment naive participants with OSA in which the adherence to therapy will be compared between TheraPAP and standard APAP. Because all participants will breathe on both therapy types and those therapy types are individually unique in feel, blinding is not possible. Participants will be chosen from a pool of patients who are PAP-naïve and who have received either a PSG (in-lab polysomnogram), split-night study (in-lab PSG and pressure titration) or home sleep study (HST) within the previous 3 months.

Upon signing an informed consent, participants will be randomly assigned to start on either the TheraPAP or APAP arms when they arrive at the office to pick up their Sefam S.Box with TheraPAP algorithms integrated. Each participant will then be given their new equipment and will be trained in proper use for both arms of the study so that they will not need to appear at the office again until the study is completed. In both the APAP and TheraPAP arms, participants will have their therapy set to 5-20 cmH2O for three nights. The pressure range will then be narrowed to ± 2 cmH2O around their 95% pressure level as assessed during the third night. This same pressure range will be used during the second arm for each patient.

Within the TheraPAP arm, participants will be set to a double Comfort Setting drop according to the following table. This drop schedule will be implemented even while the TheraPAP device is operating with automatic pressure adjustment.

Pset Drop 1 Drop 2 5.0 - 5.9 0 0 6.0 - 6.9 1 0 7.0 - 7.9 2 0 8.0 - 8.9 2 1 9.0 - 9.9 2 2 10.0 - 20.0 2 3

Participants will use their starting therapy nightly at home for 6 weeks after which time they will undergo a washout period of 1 week where no therapy will be used. Following the washout period, they will initiate another 6-week usage with the second therapy. Afterward, they will return to the office to receive their permanent equipment. Phone calls as reminders to end the first arm, start the washout period, then to start the second arm will be made.

Immediately after both arms of the study are completed, the following will occur:

* Eligibility criteria will be reviewed and confirmed
* Participants will be asked to respond to the following ESS (Epworth Sleepiness Scale) FOSQ (Functional Outcomes of Sleep Questionnaire)

During the home use period, subjects will be called at the following time points during each arm of the study. At each time point, adverse events and compliance with the device will be assessed. Subjects using the device less than an average of 5 hours per night during the first week will be contacted on a more regular basis (weekly until 5 hour per night use is achieved) to address any problems and encourage use. If patients discontinue use of the device during the home use period, they will still be encouraged to return for all testing per protocol. If a patient refuses to come in for further testing, they will be considered a lost to follow up and excluded from efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

1. AHI > 10 on a previous PSG or HST (hypopneas requiring 4% desaturation).
2. Central apneas < 25% of events
3. PLM (Periodic Limb Movements) arousal index < 15

Exclusion Criteria:

1. A female of child-bearing potential that is pregnant or intends to become pregnant.
2. Any unstable or severe medical condition of any organ system including congestive heart failure, COPD, renal failure, neuromuscular disease, etc., or at the discretion of the site Principal Investigator (PI).
3. Taking medication that may affect sleep, sleepiness, or alertness including hypnotics, sedatives, alerting agents, stimulants, anticonvulsants, etc.
4. The presence of any other sleep disorder (insomnia, periodic limb movement disorder, etc).
5. Prior therapy or treatment for OSA.
6. Chronic oxygen therapy.
7. Excessive alcohol consumption (>14 drinks/week).
8. The use of any illegal drug(s).
9. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Usage | Averaged over every night for each 6-week arm
  Number of hours for which therapy is used per night

SECONDARY OUTCOMES:
ESS Questionnaire | Filled out twice, once after completion of each 6-week arm (at week 6 and at week 13)
  Epworth Sleepiness Scale - a standard questionnaire to assess sleep quality. Scoring goes from 0 to 24 and higher scores means worsening sleepiness.
FOSQ-10 Questionnaire | Filled out twice, once after completion of each 6-week arm (at week 6 and at week 13)
  Functional Outcomes of Sleep Questionnaire - 10 - a standard questionnaire to assess sleep quality. Scoring goes from 10 to 40 and higher scores means better functional outcome.
Excess Leak or Leak | Averaged over every night for each 6-week arm
  Excess leak is patient circuit leak in excess of the normal leak required to prevent rebreathing in a CPAP device, which exits the circuit from the exhaust valve. Examples of excess leak include mask sealing leak or mouth opening. This excess leak will be averaged per night.
P95/P90 | Averaged over every night for each 6-week arm
  Standard CPAP measurement - pressure levels that eliminate breathing obstructions for at least 90% to 95% of the sleep period
AHI | Averaged over every night for each 6-week arm
  Apnea/Hypopnea Index - measure of the number of obstructive breathing events per hour experienced by the patient

CONTACTS AND LOCATIONS:
Overall Officials: William H Noah, MD, Study Director — SleepRes, LLC., Sleep Centers of Middle Tennessee, LLC
Locations (1):
- Sleep Centers of Middle Tennessee, Murfreesboro, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-05-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT06413134/Prot_000.pdf